CLINICAL TRIAL: NCT01736371
Title: Analysis of Cisatracurium Consumption in Balanced Anesthesia With 1% Sevoflurane, and With Only Sevoflurane, Using a Closed-loop Computer Controlled System Infusion.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Joomye Shehzaad, Joomye Shehzaad M.D., Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Cis-sevo-123
Record Dates: First submitted 2012-11-25; First posted 2012-11-29 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Drug Interaction Potentiation
Keywords: Sevoflurane; Cisatracurium infusion consumption; Closed loop computer control system; Recovery Index
MeSH Terms: interventions — Sevoflurane; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Total Intravenous Anesthesia (Sham Comparator): Only propofol infusion is used for maintenance of anesthesia keeping Bispectral Index (BIS) between 45-55.
  Interventions: Drug: Propofol
- 1% Sevoflurane (Active Comparator): 1% Sevoflurane with propofol infusion is used for maintenance. BIS is kept between 45-55 by adjusting propofol infusion.
  Interventions: Drug: 1% Sevoflurane
- Sevoflurane (Active Comparator): Only Sevoflurane is used for maintenance keeping BIS between 45-55
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: 1% Sevoflurane — In this group of patients, the maintenance of anesthesia is done by 1% sevoflurane + propofol infusion. Propofol infusion is adjusted according to the Bispectral Index.
  Arms: 1% Sevoflurane
Drug: Propofol — In this group the maintenance of anesthesia is maintained by only propofol infusion.
  Other Names: Total Intravenous Anesthesia
  Arms: Total Intravenous Anesthesia
Drug: Sevoflurane — In this group only sevoflurane was used for maintenance of anesthesia. the dose of sevoflurane is adjusted to maintain Bispectral Index within 45 and 55.
  Arms: Sevoflurane

SUMMARY:
The aim in this study was to quantify the difference in cisatracurium and sufentanil consumption, and its recovery period, when patients are under balanced general anesthesia with 1% sevoflurane and patients under only sevoflurane general anesthesia, using a closed loop computer control infusion. Investigators further investigated this effect on its recovery period and sufentanyl consumption.

DETAILED DESCRIPTION:
156 patients of American Society of Anesthesiologists (ASA) physical status I and II were assigned to three groups. The patients were all on schedule for elective general surgery under general anesthesia with duration of at two to four hours. All patients were induced with Etomidate (0.2mg/kg), Midazolam (0.05-0.1mg/kg), Sufentanil (0.3-0.5µg/kg) and a bolus dose of Cisatracurium (0.15mg/kg). Patients were aged between 20 and 65. The maintenance of anesthesia in each group varies as follows: Patients in Group 1 were all maintained with Total Intravenous Anesthesia, Group 2 with Sevoflurane at 1% and propofol infusion, Group 3 with only sevoflurane. Muscle paralysis is maintained using a closed-loop computer gated infusion of Cisatracurium which kept T1 <1% by giving increasing the infusion rate intra-operatively when required. Analgesia was maintained by intermittent bolus dose of 10-20 µg of Sufentanil.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 and 65.
* Patients with ASA 1 and 2.
* Patients for elective abdominal general surgery

Exclusion Criteria:

* Patients with the following diseases are excluded, since they are known to cause generalized neuromuscular weakness:

Neuromuscular junction disorders (e.g.. myasthenia gravis) Myopathies (e.g.. Muscular Dystrophies, Rhabdomyolysis) Peripheral Neuropathies (e.g. Guillain-Barre Syndrome, Polyneuropathies) Encephalopathies (Septic and Toxic-metabolic Encephalopathy) Patients with renal and liver diseases.

* Patients who are sent intubated to ICU after surgery.
* Patients refusal

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2012-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Cisatracurium consumption rate. | At the time of surgery.
  Measurements were done intraoperatively. Investigators obtained data from the closed loop computer system, from which the intra-operative consumption of cisatracurium were obtained from each patient. Data were collected only during surgery. Each patient had different cisatracurium consumption rate, and the mean consumption rate of the patients within the same group were calculated, and compared with the means from the other groups.

SECONDARY OUTCOMES:
Analysis of Means of Recovery Index. | 30 minutes post operative.
  Recovery Index was the time for the Train-Of-Four ratio (TOF) to increase from 25% to 75%. The TOF ratio was recorded every minute till it reached 90%. Time taken for each patient was from 5 to 25 minutes. Investigators compared the average recovery index of patients from each group.

OTHER OUTCOMES:
Sufentanil Consumption. | At time of surgery
  Measurements were done intraoperatively, from which the intra-operative consumption of sufentanil were obtained from each patient. Data were collected only during surgery. Investigators compared the average sufentanil consumption between between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Shehzaad Joomye, M.D., Principal Investigator — Tianjin Medical University General Hospital
Locations (1):
- Tianjin Medical University, Tianjin, China